CLINICAL TRIAL: NCT02810418
Title: A Phase Ib/II Study of Mesothelin-Targeted Immunotoxin LMB-100 Alone or in Combination With Nab-Paclitaxel in Participants With Previously Treated Metastatic and/ or Locally Advanced Pancreatic Ductal Adenocarcinoma and Mesothelin Expressing Solid Tumors
Brief Title: Mesothelin-Targeted Immunotoxin LMB-100 Alone or in Combination With Nab-Paclitaxel in People With Previously Treated Metastatic and/or Locally Advanced Pancreatic Ductal Adenocarcinoma and Mesothelin Expressing Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christine Alewine, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160128; 16-C-0128
Record Dates: First submitted 2016-06-22; First posted 2016-06-23 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Neoplasms; Pancreatic Neoplasms
Keywords: Immunotoxin; Mesothelin; Antibody-based Therapeutics; Advanced Cancer
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms | interventions — LMB-100; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (7):
- Arm A1, Dose Level 1 (Phase 1, short infusion) 100µg/kg LMB-100 (Experimental): Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 +125mg/m^2 nab-paclitaxel
  Dose level 1 (DL1) Maximum tolerated dose (MTD) determination in patients with pancreatic cancer receiving short infusion LMB-100+nabpaclitaxel
  Interventions: Drug: LMB-100; Drug: Nab-Paclitaxel
- Arm A1, Dose Level-1 (Phase 1, short infusion) 65µg/kg LMB-100 (Experimental): Arm A1, DL-1, Ph I Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel
  Interventions: Drug: LMB-100; Drug: Nab-Paclitaxel
- Arm A2 (Phase 2, short infusion) 65µg/kg LMB-100 (Experimental): Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel
  Efficacy determination in patients with pancreatic cancer receiving short infusion LMB-100 + nabpaclitaxel
  Interventions: Drug: LMB-100; Drug: Nab-Paclitaxel
- Arm B1, Dose Level 2 Phase I (Continuous infusion single agent lead-in) (Experimental): Arm B1, DL2, 48-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 Maximum tolerated dose (MTD) determination in patients with pancreatic cancer receiving continuous infusion LMB-100 as single agent
  Interventions: Drug: LMB-100; Device: Mesothelin Expression
- Arm B1, Dose Level 1 Phase I (Continuous infusion single agent lead-in) (Experimental): Arm B1, DL1, 48-hr Continuous Infusion Single Agent Lead-in 65µg/kg/day LMB-100
  Interventions: Drug: LMB-100; Device: Mesothelin Expression
- Arm B1, Dose Level 3R Phase I (Continuous infusion single agent lead-in) (Experimental): Arm B1, DL3R, 24-hr Continuous Infusion Single Agent Lead-in 100µg/kg LMB-100
  Interventions: Drug: LMB-100; Device: Mesothelin Expression
- Arm B2 Phase I (continuous infusion combination therapy) (Experimental): Subjects with pancreatic cancer receiving continuous infusion LMB-100 combination therapy
  Interventions: Drug: LMB-100; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: LMB-100 — Arms A1 and A2 (short infusion): Administered intravenously (IV) on days 1, 3 and 5 of a 21 day cycle for a maximum of 2 cycles Arm B1 (continuous infusion): Administered IV for 24, 48, 72 or 96 hours continuously on the first 1 - 4 days or 24 hour infusions on days 1 and 4 (depending on dose level) of each 21 day cycle for a maximum of 2 cycles. Arm B2 (continuous infusion): Administered IV for 24,48, 72 or 96 hours continuously on the first 1 - 4 days or 24 hour infusions on days 1 and 4 (depending on dose level) of each 14 day cycle for a maximum of 3 cycles.
Drug: Nab-Paclitaxel — Administered intravenously (IV) on days 1 and for Arms A1, A2 and B1 on day 8 of each 14-21 day cycle for a maximum of 2 (Arms A1, A2 and B1) or 3 (Arm B2) cycles
  Other Names: Abraxane
  Arms: Arm A1, Dose Level 1 (Phase 1, short infusion) 100µg/kg LMB-100; Arm A1, Dose Level-1 (Phase 1, short infusion) 65µg/kg LMB-100; Arm A2 (Phase 2, short infusion) 65µg/kg LMB-100; Arm B2 Phase I (continuous infusion combination therapy)
Device: Mesothelin Expression — Research blood test for Arm B1 eligibility
  Arms: Arm B1, Dose Level 1 Phase I (Continuous infusion single agent lead-in); Arm B1, Dose Level 2 Phase I (Continuous infusion single agent lead-in); Arm B1, Dose Level 3R Phase I (Continuous infusion single agent lead-in)
Drug: LMB-100 — A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.
  Arms: Arm B1, Dose Level 2 Phase I (Continuous infusion single agent lead-in); Arm B1, Dose Level 3R Phase I (Continuous infusion single agent lead-in); Arm B2 Phase I (continuous infusion combination therapy)

SUMMARY:
Background:

LMB-100 is a man-made protein designed to kill cancer cells. LMB-100 targets a cancer marker called mesothelin. Mesothelin is found on the surface of many different tumors, including pancreatic cancer, but is made by a very small number of normal tissues. Other cancers that make mesothelin include mesothelioma, cholangiocarcinoma, thymic carcinoma, ovarian, lung, gastric, endometrial, cervical, and ampullary cancers. After binding to the mesothelin on tumors, LMB-100 can attack and kill cancer cells. Researchers want to see how well it works when given with and without nab-paclitaxel, a drug which treats pancreatic cancer.

Objectives:

Arm A- To find a safe dose of LMB-100 with a fixed standard dose of nab-paclitaxel in people with advanced pancreatic cancer. To see how well the combination of the two drugs reduce tumor size.

Arm B- To find a safe dose of LMB-100 when it is given as a continuous infusion over several days.

Eligibility:

Arm A- Adults age 18 and older with advanced pancreatic cancer that has worsened after anti-cancer therapy.

Arm B- Adults age 18 and older with advanced pancreatic cancer, mesothelioma or other solid tumor that makes mesothelin that has worsened after anti-cancer therapy

Design:

Participants will be screened with medical history and physical exam. They will give blood, urine, and tissue samples. They will have scans and x-rays.

During each 21-day cycle:

* For Arm A

  * Participants will get LMB-100 by an intravenous (IV) catheter on days 1, 3, and 5. This is a tube inserted in a vein, usually in the arm.
  * Participants will get nab-paclitaxel by IV on days 1 and 8.
* For Arm B

  * Participants will get LMB-100 by an IV catheter as a continuous infusion beginning on day 1 and continuing for 2-4 days
  * Some participants will also get nab-paclitaxel by IV on days 1 and 8.

All participants will get this combination for up to 2 cycles or until their disease worsens or they have intolerable side effects.

Participants will have blood and urine tests and scans throughout the study.

Participants will have a safety follow-up visit 3-6 weeks after treatment ends. If their disease remains stable or improves, they will be scanned every 6 weeks until their disease gets worse. Even if their disease gets worse, they or their doctor will be called to talk about their cancer status....

DETAILED DESCRIPTION:
Background:

* Pancreatic cancer is the fourth most common cause of cancer death in the United States, claiming more than 40,000 lives each year.
* Incidence nearly equals mortality with just 6% of participants living five years beyond their diagnosis. Most patients are diagnosed at an advanced stage, but even patients with early stage disease have a long term survival of less than 20%.
* Mesothelin is specifically a marker of adenocarcinoma in the human disease and is not expressed in preceding pre-malignant stages of tumor development
* Expression of mesothelin in pancreatic ductal adenocarcinoma (PDA) has been examined in several published studies and ranges from 86 to 100%
* Recombinant immunotoxins (RITs) are antibody-based therapeutics that carry a toxin payload. RITs that target mesothelin contain a genetically engineered variant of Pseudomonas exotoxin A (PE) in which the native cell-binding domain of PE is replaced by the mesothelin-binding antibody fragment. SS1P was the first mesothelin-targeted RIT tested in patients.
* LMB-100 contains a newly engineered PE fragment that has improved activity against most pancreatic cancer cell lines in vitro, and is also much less toxic than SS1P in preclinical models. The new PE contains modifications specifically designed to reduce immunogenicity of the molecule.
* Pre-administration of paclitaxel with SS1P was demonstrated to increase the amount of immunotoxin internalized by tumor cells and to reduce levels of shed mesothelin in the intra-tumoral environment so that more immunotoxin could bind tumor cells. The effect is even more pronounced with NAB-paclitaxel in a pancreatic cancer model.
* Initial clinical testing of LMB-100 was performed by Roche in a multi-center international first in human trial (NCT02317419). The agent was well tolerated and appeared to have decreased immunogenicity compared to SS1P based on preliminary results.
* In initial and subsequent clinical testing, LMB-100 was found to have half-life of approximately 60 mins. This is shorter then that measured for previous RITs used in the clinical setting.

Primary Objectives:

* Arm A1 (Phase I, short infusion):

  --To determine the maximum tolerated dose of short infusion LMB-100 in combination nab-paclitaxel chemotherapy in participants with advanced pancreatic cancer
* Arm B1(Continuous infusion single agent lead-in):

  --To determine the maximum tolerated dose of LMB-100 given in a continuous infusion format over 24 - 96 hours to patients with advanced solid tumors that express mesothelin
* Arm B2 (Continuous infusion combination therapy)

  --Establish a tolerated dose of LMB-100 given by continuous infusion in combination with nab-paclitaxel chemotherapy in participants with advanced pancreatic cancer
* Arm A2 (Phase II, short infusion):

  * To determine the objective response rate (Partial Response (PR)+Complete Response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria of short infusion LMB-100 in combination with nab-paclitaxel chemotherapy in participants with advanced pancreatic cancer

Eligibility:

* Age greater than or equal to18 years
* Histologically confirmed recurrent, metastatic and/or advanced pancreatic ductal adenocarcinoma (Except for Arm B1 [B Single Agent Lead-in])
* For Arm B1 (Single Agent Lead-in), ONLY: Histologically confirmed solid tumor malignancy for which no curative therapy exists with at least 25% of tumor cells expressing mesothelin as determined by National Cancer Institute (NCI) Laboratory of Pathology. Determination can be made using archival tumor tissue or fresh biopsy.
* Treatment must include at least one prior chemotherapy regimen
* No nab-paclitaxel or paclitaxel treatment in the last four months (Except for Arm B1 [Single Agent Lead-in])
* Adequate organ function
* Participants with human immunodeficiency virus (HIV), active hepatitis B virus (HBV) or hepatitis C virus (HCV) infections are eligible only for the Arm B1 (Single Agent Lead-in)

Design:

* This study is a Phase I/II open label study to assess the safety and efficacy of LMB-100 in combination with the standard of care agent nab-paclitaxel in participants metastatic and/or locally advanced pancreatic ductal adenocarcinoma
* Subjects will be treated for up to 2 cycles
* In Arm A1 (Phase I, short infusion) of the study, up to 3 dose levels will be evaluated. LMB-100 will be administered on days 1, 3 and 5 of a 21 day cycle and nab-paclitaxel will be administered on days 1 and 8
* Arm A2 (Phase II, short infusion), up to 20 evaluable participants (including those treated at the short infusion maximum tolerated dose (MTD) in the phase I study) will be enrolled.
* Arm B1 (Continuous infusion single Agent Lead-in), escalating doses of single agent LMB-100 will be administered. The study drug will be given as a continuous infusion for the 1, 2, 3, or 4 days of a 21-day cycle.
* Arm B2 (Continuous infusion, combination therapy) will be initiated after completion of both Arm A1 and Arm B1 Single Agent Lead-in. It will test a single dose level of LMB-100 based on data from the Lead-in given in combination with nab-paclitaxel. LMB-100 will be given as a continuous infusion for the 1, 2, 3 or 4 days of a 21-day cycle. Nabpaclitaxel will be given on Day 1 and Day 8.
* The Arm A2 (Phase II, short infusion) portion of the study will be conducted in a Simon Minimax two stage phase II design. The first stage will enroll 13 evaluable participants, including the six participants treated at the short infusion MTD from phase I. If 1 or more has a response, then accrual would continue until a total of 20 evaluable participants have been enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:
* For participants who will be receiving nab-paclitaxel (all arms except Phase I Arm B Single Agent Lead-in)

  * Histologically confirmed recurrent, advanced or metastatic pancreatic ductal adenocarcinoma as determined by National Cancer Institute (NCI) Laboratory of Pathology.
  * No treatment with paclitaxel or nab-paclitaxel within 4 months prior to initiation of study therapy
  * Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
  * Adequate hematological function: neutrophil count of greater than or equal to 1.0 x 10(9) cells/L, platelet count of greater than or equal to 95,000/microliters, hemoglobin greater than or equal to 9 g/dL
  * Measurable disease as per the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria v 1.1
  * For participants who will NOT receive nab-paclitaxel (Arm B1 Single Agent Lead-in only)
  * Histologically confirmed solid tumor malignancy for which no curative therapy exists with at least 25% of tumor cells expressing mesothelin as determined by NCI Laboratory of Pathology. Determination can be made using archival tumor tissue or fresh biopsy. Subjects with epithelioid mesothelioma and pancreatic adenocarcinoma are automatically eligible and are not required to have this test.
  * ECOG performance status (PS) 0-2.
  * Adequate hematological function: neutrophil count of greater than or equal to 1.0 x 10(9) cells/L, platelet count of greater than or equal to 85,000/microliters, hemoglobin greater than or equal to 8.5 g/dL
  * Measurable and/or evaluable disease as per the RECIST Criteria v 1.1
* For all arms of the protocol

  * Participants must have received at least one prior chemotherapy regimen for their disease.
  * Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of LMB-100 in combination with nab-paclitaxel in persons <18 years of age, children are excluded from this study.
  * Participants must be more than 14 days removed from most recent minor surgical procedure (such as biliary stenting), 28 days from most recent major surgical procedure, 14 days removed from most recent radiation therapy, chemotherapy or experimental drug treatment with published half-life known to be 72 hours or less and 28 days removed from last experimental drug treatment with unpublished or half-life greater than 72 hours.
  * All acute toxic effects of any prior radiotherapy, chemotherapy, experimental drug treatment or surgical procedure must have resolved to Grade less than or equal to 1, except alopecia (any grade) and peripheral neuropathy.
  * Serum albumin greater than or equal to 2.5 mg/dL without intravenous supplementation
  * Adequate liver function: Bilirubin, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN). AST and ALT up to 5x ULN is permitted for patients with liver metastases.
  * Adequate renal function: creatinine clearance greater than or equal to 50 mL/min.
  * Must have left ventricular ejection fraction > 50%
  * Must have an ambulatory oxygen saturation of > 88% on room air
  * The effects of LMB-100 alone or in combination with nab-paclitaxel on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry until 3 months the last dose of study therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Exclusion criteria for all study arms

  * Known or clinically suspected central nervous system (CNS) 2.1.2.1 primary tumors or metastases including leptomeningeal metastases. History or clinical evidence of CNS metastases unless they have been previously treated, are asymptomatic, and have had no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days.
  * Evidence of significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results, including significant pulmonary disease other than that related to the primary cancer, uncontrolled diabetes mellitus, and/or significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, unstable angina, or clinically significant pericardial effusion)
  * Any known diagnoses, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition (other than pancreatic adenocarcinoma) that would contraindicate the use of an investigational drug, interfere with tumor measurement or lead to an expected life expectancy of less than 6 months as judged by the investigator
  * Active or uncontrolled infections.
  * Live attenuated vaccinations within 14 days prior to treatment
  * Dementia or altered mental status that would prohibit informed consent
  * Pregnant women are excluded from this study because the effects of LMB-100 on the developing fetus are unknown and may have the potential to cause teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LMB-100, breastfeeding should be discontinued if the mother is treated with LMB-100. These potential risks may also apply to other agents used in this study.
  * Known hypersensitivity to any of the components of LMB-100
  * Baseline corrected QT interval by Fridericia (QTcF) interval of > 470 ms, participants with baseline resting bradycardia < 45 beats per minute, or baseline resting tachycardia> 100 beats per minute.
* Exclusion criteria specific to patients who will be receiving nab-paclitaxel (all arms except Arm B1 Single Agent Lead-in)

  * Participants with contra-indication and/or history of severe hypersensitivity reactions to nab-paclitaxel
  * Participants with baseline peripheral neuropathy greater than grade 2
  * Human immunodeficiency virus (HIV) or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection due to risk of progression while receiving immunosuppressive chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine C Alewine, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pegna GJ, Lee MJ, Peer CJ, Ahmad MI, Venzon DJ, Yu Y, Yuno A, Steinberg SM, Cao L, Figg WD, Donahue RN, Hassan R, Pastan I, Trepel JB, Alewine C. Systemic immune changes accompany combination treatment with immunotoxin LMB-100 and nab-paclitaxel. Cancer Med. 2023 Feb;12(4):4236-4249. doi: 10.1002/cam4.5290. Epub 2022 Oct 8. PMID 36208017
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0128.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100: Arm A1, DL1, Ph I Short Infusion 100µg/kg LMB-100 +125mg/m^2 nab-paclitaxel LMB-100 (short infusion): Administered intravenously (IV) on days 1, 3 and 5 of a 21 day cycle for a maximum of 2 cycles;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on days 1, and 8 of each 21 day cycle for a maximum of 2 cycles
- Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100: Arm A1, DL-1, Ph I Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel
  LMB-100 (short infusion): Administered intravenously (IV) on days 1, 3 and 5 of a 21 day cycle for a maximum of 2 cycles;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on days 1, and 8 of each 21 day cycle for a maximum of 2 cycles
- Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100: Arm A2, Ph 2 Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel
  LMB-100 (short infusion): Administered intravenously (IV) on days 1, 3 and 5 of a 21 day cycle for a maximum of 2 cycles;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on days 1, and 8 of each 21 day cycle for a maximum of 2 cycles
- Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in: Arm B1, DL2, 48-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered intravenously (IV)for 48 hours continuously on the first 1 - 2 days of each 21 day cycle for a maximum of 2 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion
- Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in: Arm B1, DL1, 48-hr Continuous Infusion Single Agent Lead-in 65µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered intravenously (IV) for 48 hours continuously on the first 1 - 2 days of each 21 day cycle for a maximum of 2 cycles
- Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in: Arm B1, DL3R, 24-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered IV for 24 hours continuously starting on days 1 and 4 of each 21 day cycle for a maximum of 2 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.
- Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg: Arm B2, 24-hr Continuous Infusion Combo Therapy 100µg/kg/day LMB-100+125mg/m^ nab-paclitaxel Arms B2 (continuous infusion LMB-100): Administered intravenously (IV) for 24 hours continuously starting on day 1 of each 14 day cycle for a maximum of 3 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on day 1of each 14 day cycle for a maximum of 3 cycles
Period: Arm A Dose Escalation
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 | Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
Started | 6 | 8 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 7 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 | Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
Started | 0 | 8 | 6 | 0 | 0 | 0 | 0
Completed | 0 | 7 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Arm B Dose Escalation
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 | Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
Started | 0 | 0 | 0 | 6 | 3 | 6 | 0
Completed | 0 | 0 | 0 | 6 | 2 | 4 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2 | 0
Period: Arm B Combination Therapy
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 | Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in: Arm B1, DL1, 48-hr Continuous Infusion Single Agent Lead-in 65µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered IV for 48 hours continuously on the first 1 - 4 days of each 21 day cycle for a maximum of 2 cycles
- Total: Total of all reporting groups
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 | Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg | Total
Number analyzed (Participants) | 6 | 8 | 6 | 6 | 3 | 6 | 5 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 2 | 4 | 3 | 3 | 2 | 25
  >=65 years | 0 | 3 | 4 | 2 | 0 | 3 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (7.6) | 61.0 (7.7) | 69.9 (8.5) | 47.0 (12.5) | 59.2 (12.3) | 62.8 (7.9) | 66.8 (10.4) | 61.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 2 | 2 | 1 | 3 | 18
  Male | 4 | 4 | 2 | 4 | 1 | 5 | 2 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 8 | 5 | 6 | 3 | 6 | 2 | 36
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 4
  White | 6 | 7 | 6 | 4 | 1 | 4 | 4 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 6 | 6 | 3 | 6 | 5 | 40
Number of Participants with Prior Therapies [Count of Participants; unit: Participants]
  Whipple | 2 | 5 | 4 | 2 | 1 | 3 | 3 | 20
  Radiation | 5 | 4 | 5 | 4 | 2 | 2 | 4 | 26
  Prior nab-paclitaxel | 1 | 3 | 2 | 5 | 1 | 5 | 3 | 20
Number of Participants with Sites of Disease [Count of Participants; unit: Participants]
  Liver | 4 | 5 | 4 | 3 | 3 | 4 | 1 | 24
  Lung | 2 | 5 | 4 | 3 | 3 | 3 | 3 | 23
  Other | 2 | 3 | 6 | 5 | 3 | 3 | 3 | 25
  Ascites | 1 | 0 | 2 | 2 | 1 | 2 | 0 | 8
Participants Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — ECOG 0 is normal activity; 1 is symptoms, but ambulatory; and 2 is in bed<50% of the time.
  Participants
    0 | 2 | 4 | 3 | 2 | 0 | 1 | 2 | 14
    1 | 4 | 4 | 3 | 4 | 1 | 5 | 3 | 24
    2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Baseline CA 19-9 [Number; unit: Unit/mL] — CA 19-9 serum tumor marker normal values is between 0 and 37 U/mL. High values can indicate pancreatic cancer.
  Unit/mL
    Patient 1 | 404.7 | 0 | 0 | 0 | 0 | 0 | 0 | 404.7
    Patient 2 | 10650 | 0 | 0 | 0 | 0 | 0 | 0 | 10650
    Patient 3 | 248800 | 0 | 0 | 0 | 0 | 0 | 0 | 248800
    Patient 4 | 27.8 | 0 | 0 | 0 | 0 | 0 | 0 | 27.8
    Patient 5 | 7081 | 0 | 0 | 0 | 0 | 0 | 0 | 7081
    Patient 6 | 0 | 0 | 0 | 0 | 123 | 0 | 0 | 123
    Patient 7 | 1277 | 0 | 0 | 0 | 0 | 0 | 0 | 1277
    Patient 8 | 0 | 0 | 0 | 0 | 94210 | 0 | 0 | 94210
    Patient 9 | 0 | 0 | 0 | 0 | 1500 | 0 | 0 | 1500
    Patient 10 | 0 | 10106 | 0 | 0 | 0 | 0 | 0 | 10106
    Patient 11 | 0 | 0 | 0 | 13.2 | 0 | 0 | 0 | 13.2
    Patient 12 | 0 | 25180 | 0 | 0 | 0 | 0 | 0 | 25180
    Patient 13 | 0 | 0 | 0 | 14.8 | 0 | 0 | 0 | 14.8
    Patient 14 | 0 | 0 | 0 | 911.3 | 0 | 0 | 0 | 911.3
    Patient 15 | 0 | 88.4 | 0 | 0 | 0 | 0 | 0 | 88.4
    Patient 16 | 0 | 0 | 0 | 284.7 | 0 | 0 | 0 | 284.7
    Patient 17 | 0 | 302.6 | 0 | 0 | 0 | 0 | 0 | 302.6
    Patient 18 | 0 | 4206 | 0 | 0 | 0 | 0 | 0 | 4206
    Patient 19 | 0 | 0 | 0 | 93.7 | 0 | 0 | 0 | 93.7
    Patient 20 | 0 | 4482 | 0 | 0 | 0 | 0 | 0 | 4482
    Patient 21 | 0 | 0 | 0 | 142.9 | 0 | 0 | 0 | 142.9
    Patient 22 | 0 | 0 | 0 | 0 | 0 | 446.6 | 0 | 446.6
    Patient 23 | 0 | 0 | 0 | 0 | 0 | 389.5 | 0 | 389.5
    Patient 24 | 0 | 0 | 0 | 0 | 0 | 156.8 | 0 | 156.8
    Patient 25 | 0 | 13348 | 0 | 0 | 0 | 0 | 0 | 13348
    Patient 26 | 0 | 0 | 0 | 0 | 0 | 9254 | 0 | 9254
    Patient 27 | 0 | 0 | 0 | 0 | 0 | 138.3 | 0 | 138.3
    Patient 28 | 0 | 0.6 | 0 | 0 | 0 | 0 | 0 | 0.6
    Patient 29 | 0 | 0 | 0 | 0 | 0 | 9571 | 0 | 9571
    Patient 30 | 0 | 0 | 2077 | 0 | 0 | 0 | 0 | 2077
    Patient 31 | 0 | 0 | 0 | 0 | 0 | 0 | 3424 | 3424
    Patient 32 | 0 | 0 | 0 | 0 | 0 | 0 | 9326 | 9326
    Patient 33 | 0 | 0 | 0 | 0 | 0 | 0 | 760 | 760
    Patient 34 | 0 | 0 | 0 | 0 | 0 | 0 | 3297 | 3297
    Patient 35 | 0 | 0 | 0 | 0 | 0 | 0 | 6345 | 6345
    Patient 36 | 0 | 0 | 2966 | 0 | 0 | 0 | 0 | 2966
    Patient 37 | 0 | 0 | 99.8 | 0 | 0 | 0 | 0 | 99.8
    Patient 38 | 0 | 0 | 1340 | 0 | 0 | 0 | 0 | 1340
    Patient 39 | 0 | 0 | 31440 | 0 | 0 | 0 | 0 | 31440
    Patient 40 | 0 | 0 | 3857 | 0 | 0 | 0 | 0 | 3857

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR) (Partial Responses + Complete Responses) in Phase 2 Subjects of Short Infusion LMB-100+ Nab-paclitaxel
Description: OR is defined as partial responses + complete response in participants in the phase 2 Arm A portion of the study assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Complete Response is a disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters
Time Frame: Approximately 6 weeks after the start of treatment and continuing every 6 weeks until progression or start of a new treatment, up to 1 year
Measure: Count of Participants; unit: Participants
Groups:
- All Participants in Arm A1 DL-1 and Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100: All participants in Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 Arm A1, DL-1, Ph I Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel LMB-100 (short infusion): Administered intravenously (IV) on days 1, 3 and 5 of a 21 day cycle for a maximum of 2 cycles;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on days 1, and 8 of each 21 day cycle for a maximum of 2 cycles AND Arm A2, Ph 2 Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel LMB-100 (short infusion): Administered intravenously (IV) on days 1, 3 and 5 of a 21 day cycle for a maximum of 2 cycles;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on days 1, and 8 of each 21 day cycle for a maximum of 2 cycles
Arm/Group | All Participants in Arm A1 DL-1 and Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100
Number analyzed (Participants) | 14
Participants | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Short Infusion LMB-100 + Nab Paclitaxel
Description: MTD is defined as the highest dose tolerated without exceeding a pre-set number of adverse events in Phase 1, Arm A.
Time Frame: 21 days after LMB-100 is administered (end of cycle 1)
Measure: Number; unit: µg/kg
Groups:
- All Participants in Arm A1, Dose Level-1, and Arm A1 Dose Level 1 Phase I Short Infusion: All participants in Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 Arm A1, DL-1, Ph I Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel LMB-100 (short infusion): Administered intravenously (IV) on days 1, 3 and 5 of a 21 day cycle for a maximum of 2 cycles;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on days 1, and 8 of each 21 day cycle for a maximum of 2 cycles AND Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 Arm A1, DL1, Ph I Short Infusion 100µg/kg LMB-100 +125mg/m^2 nab-paclitaxel LMB-100 (short infusion): Administered intravenously (IV) on days 1, 3 and 5 of a 21 day cycle for a maximum of 2 cycles;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on days 1, and 8 of each 21 day cycle for a maximum of 2 cycles
Arm/Group | All Participants in Arm A1, Dose Level-1, and Arm A1 Dose Level 1 Phase I Short Infusion
Number analyzed (Participants) | 14
µg/kg | 65

3. Primary Outcome: Maximum Tolerated Dose (MTD) of Continuous Infusion LMB-100
Description: MTD is defined as the highest dose tolerated without exceeding a pre-set number of adverse events in Phase 1, 1 Arm B, single agent lead-in
Time Frame: 21 days after LMB-100 is administered (end of cycle 1)
Population: Arm B2, Phase I, 24-hour continuous infusion combination therapy is not reported here because MTD was only assessed in the Phase I, Arm B single agent lead-in Arm/Groups.
  Please note: Dose 100 (µg/kg/day), for duration (24 Hours), schedule Days 1 & 4, preceded by a 40 mcg/kg loading dose over 30 minutes, was determined to be the preferred schedule.
Measure: Number; unit: Dose (µg/kg)
Groups:
- All Participants in Arm B1 DL2 and Arm B1 DL 1 and Arm B1 DL3R Phase I 48-hr Continuous Infusion: All participants in Arm B1, DL2, 48-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered intravenously (IV)for 48 hours continuously on the first 1 - 2 days of each 21 day cycle for a maximum of 2 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.
  AND Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in Arm B1, DL1, 48-hr Continuous Infusion Single Agent Lead-in 65µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered IV for 48 hours continuously on the first 1 - 4 days of each 21 day cycle for a maximum of 2 cycles AND Arm B1, DL3R, 24-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered IV for 24 hours continuously starting on days 1 and 4 of each 21 day cycle for a maximum of 2 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.
Arm/Group | All Participants in Arm B1 DL2 and Arm B1 DL 1 and Arm B1 DL3R Phase I 48-hr Continuous Infusion
Number analyzed (Participants) | 15
Dose (µg/kg) | 100

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is the average time from treatment initiation to disease progression or death. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. And the appearance of one or more new lesions.
Time Frame: Time from treatment initiation to disease progression or death, an average of 1 year.
Population: It was specified in the protocol that patients enrolled in Arm A1 who received the maximum tolerated dose (MTD) should be included for PFS endpoint analysis of Arm A2 data. Therefore, 8 (Arm A1, DL-1) + 6 (Arm A2) = 14 patients were included in the Arm 2 PFS analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in: Arm B1, DL1, 48-hr Continuous Infusion Single Agent Lead-in 65µg/kg LMB-100
  (continuous infusion LMB-100 as a single agent): Administered intravenously (IV) for 48 hours continuously on the first 1 - 4 days of each 21 day cycle for a maximum of 2 cycles
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 | Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
Number analyzed (Participants) | 6 | 8 | 14 | 3 | 6 | 6 | 5
Months | NA [NA to NA] — We are unable to calculate PFS of the regimen in any arm because multiple participants with stable disease immediately went on to receive other treatments following their planned 2 cycles of LMB-100. | NA [NA to NA] — We are unable to calculate PFS of the regimen in any arm because multiple participants with stable disease immediately went on to receive other treatments following their planned 2 cycles of LMB-100. | NA [NA to NA] — We are unable to calculate PFS of the regimen in any arm because multiple participants with stable disease immediately went on to receive other treatments following their planned 2 cycles of LMB-100. | NA [NA to NA] — We are unable to calculate PFS of the regimen in any arm because multiple participants with stable disease immediately went on to receive other treatments following their planned 2 cycles of LMB-100. | NA [NA to NA] — We are unable to calculate PFS of the regimen in any arm because multiple participants with stable disease immediately went on to receive other treatments following their planned 2 cycles of LMB-100. | NA [NA to NA] — We are unable to calculate PFS of the regimen in any arm because multiple participants with stable disease immediately went on to receive other treatments following their planned 2 cycles of LMB-100. | NA [NA to NA] — We are unable to calculate PFS of the regimen in any arm because multiple participants with stable disease immediately went on to receive other treatments following their planned 2 cycles of LMB-100.

5. Secondary Outcome: Overall Survival (OS)
Description: OS is the average time from treatment initiation to death.
Time Frame: Time from treatment initiation to death, up to 1-2 years.
Population: Arm/Groups A1 and B1 are not separated per Arm/Group because the breakdown by individual treatment group within each arm results in numbers that are so small that the data becomes virtually useless. Patients enrolled in A1 who were treated at the maximum tolerated dose (MTD) and meet the eligibility requirement for A2 are also counted toward the A2 endpoints as per protocol.
Measure: Median (Standard Deviation); unit: Days
Groups:
- All Participants in Arm A1 Phase I Short Infusion: All participants in Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg, and Arm A1, DL-1, Ph I Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel
- All Participants in Arm A2, Phase 2 Short Infusion: All participants in Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel
- All Participants in Arm B1 Phase I Continuous Infusion: All participants in Arm B1, DL2, 48-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered intravenously (IV)for 48 hours continuously on the first 1 - 2 days of each 21 day cycle for a maximum of 2 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion AND Arm B1, DL1, 48-hr Continuous Infusion Single Agent Lead-in 65µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered intravenously (IV) for 48 hours continuously on the first 1 - 2 days of each 21 day cycle for a maximum of 2 cycles AND Arm B1, DL3R, 24-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered IV for 24 hours continuously starting on days 1 and 4 of each 21 day cycle for a maximum of 2 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.
- All Participants in Arm B2, Phase I 24-hr Continuous Infusion Combo: All participants in Arm B2, 24-hr Continuous Infusion Combo Therapy 100µg/kg/day LMB-100+125mg/m^ nab-paclitaxel Arms B2 (continuous infusion LMB-100): Administered intravenously (IV) for 24 hours continuously starting on day 1 of each 14 day cycle for a maximum of 3 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on day 1of each 14 day cycle for a maximum of 3 cycles
Arm/Group | All Participants in Arm A1 Phase I Short Infusion | All Participants in Arm A2, Phase 2 Short Infusion | All Participants in Arm B1 Phase I Continuous Infusion | All Participants in Arm B2, Phase I 24-hr Continuous Infusion Combo
Number analyzed (Participants) | 14 | 14 | 15 | 5
Days | 202 (332) | 160 (196) | 89 (124) | 167 (348)

6. Secondary Outcome: Proportion of Participants Disease Control Rate (DCR) at End of Treatment (EOT)
Description: DCR is the proportion of participants with stable disease, partial response or complete response at end of treatment. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Complete Response is disappearance of all target lesions. Stable disease is neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: up to 3 months
Population: It was planned that this outcome measure would be reported by Arm and not by individual dose levels within each arm. Pts enrolled in A1 who were treated at the max.tolerated dose and meet the eligibility requirement for A2 are also counted toward the A2 endpoints as per protocol. We are unable to calculate DCR at 4 mos because many pts with stable disease immediately went on to receive other therapies following completion of scheduled 2-3 cycles of LMB-100. Therefore,we are reporting DCR at EOT.
Measure: Number; unit: Proportion of participants
Groups:
- All Participants in Arm A2 Phase 2 Short Infusion: All participants in Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel
- All Participants in Arm B1 Phase I Continuous Infusion: All participants in Arm B1, DL2, 48-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered intravenously (IV)for 48 hours continuously on the first 1 - 2 days of each 21 day cycle for a maximum of 2 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.
  AND Arm B1, DL1, 48-hr Continuous Infusion Single Agent Lead-in 65µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered intravenously (IV) for 48 hours continuously on the first 1 - 2 days of each 21 day cycle for a maximum of 2 cycles AND Arm B1, DL3R, 24-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered IV for 24 hours continuously starting on days 1 and 4 of each 21 day cycle for a maximum of 2 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.
Arm/Group | All Participants in Arm A1 Phase I Short Infusion | All Participants in Arm A2 Phase 2 Short Infusion | All Participants in Arm B1 Phase I Continuous Infusion | All Participants in Arm B2, Phase I 24-hr Continuous Infusion Combo
Number analyzed (Participants) | 14 | 14 | 15 | 5
Proportion of participants
  Partial Response | 0.07 | 0.07 | 0 | 0
  Complete Response | 0 | 0 | 0 | 0
  Stable Disease | 0.71 | 0.5 | 0.27 | 0.4
  Progressive Disease | 0.21 | 0.36 | 0.60 | 2
  Not Evaluable | 0 | 0.07 | 0.13 | 1

7. Secondary Outcome: Number of Participants With an Objective Response (OR) (Partial Responses + Complete Responses) in Phase 1 Arm A1
Description: OR is defined as partial response + complete response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Complete Response is a disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters
Time Frame: Approximately 6 weeks after the start of treatment and continuing every 6 weeks until progression or start of a new treatment up to 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100
Number analyzed (Participants) | 6 | 8
Participants | 0 | 1

8. Secondary Outcome: Number of Participants With an Objective Response (OR) (Partial Response + Complete Response) in Phase 1, Arm B
Description: OR is defined as partial responses + complete response in participants in the phase 1 Arm B portion of the study assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Complete Response is a disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in: Arm B1, DL1, 48-hr Continuous Infusion Single Agent Lead-in 65µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered intravenously (IV) for 48 hours continuously on the first 1 - 4 days of each 21 day cycle for a maximum of 2 cycles
Arm/Group | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in
Number analyzed (Participants) | 6 | 3 | 6
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Adverse Events Attributed to LMB-100
Description: Grade 1-4 adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v4.0 observed in subjects with pancreatic cancer. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe or medically significant. Grade 4 is life-threatening consequences.
Time Frame: Date treatment consent signed to date off study, approx. 11 mos, 8 days for A1DL1; 20 mos, 9 days for A1DL-1; 10 mos, 17 days for A2; 2 mos, 16 days for B1DL1; 14 mos, 30 days for B1DL2; 5 mos, 1 day for B2; and 4 mos, 15 days for B1DL3R.
Population: No B2 grade 1, 3, and 4; B1 DL1 grade 1, 3, and 4; B1 DL2 grade 1; and B1 DL3R grade 1, 3, and 4 adverse events.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A1, Dose Level 1 Phase I Grade 1; Arm A1, Dose Level-1 Phase I Grade 1; Arm A2, Phase 2 Grade 1: Grade 1 mild adverse events.
- Arm A1, Dose Level 1 Phase I Grade 2; Arm A1, Dose Level-1 Phase I Grade 2; Arm A2, Phase 2 Grade 2; Arm B1, Dose Level 2 Phase I Grade 2; Arm B1, Dose Level 1 Phase I Grade 2; Arm B1, Dose Level 3R Phase I Grade 2; Arm B2 Phase I Grade 2: Grade 2 moderate adverse events.
- Arm A1, Dose Level 1 Phase I Grade 3; Arm A1, Dose Level-1 Phase I Grade 3; Arm A2, Phase 2 Grade 3; Arm B1, Dose Level 2 Phase I Grade 3: Grade 3 severe or medically significant adverse events.
- Arm A1, Dose Level-1 Phase I Grade 4; Arm A2, Phase 2 Grade 4; Arm B1, Dose Level 2 Phase I Grade 4: Grade 4 life-threatening adverse events.
Arm/Group | Arm A1, Dose Level 1 Phase I Grade 1 | Arm A1, Dose Level 1 Phase I Grade 2 | Arm A1, Dose Level 1 Phase I Grade 3 | Arm A1, Dose Level-1 Phase I Grade 1 | Arm A1, Dose Level-1 Phase I Grade 2 | Arm A1, Dose Level-1 Phase I Grade 3 | Arm A1, Dose Level-1 Phase I Grade 4 | Arm A2, Phase 2 Grade 2 | Arm A2, Phase 2 Grade 1 | Arm A2, Phase 2 Grade 3 | Arm A2, Phase 2 Grade 4 | Arm B1, Dose Level 2 Phase I Grade 2 | Arm B1, Dose Level 2 Phase I Grade 3 | Arm B1, Dose Level 2 Phase I Grade 4 | Arm B1, Dose Level 1 Phase I Grade 2 | Arm B1, Dose Level 3R Phase I Grade 2 | Arm B2 Phase I Grade 2
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 5
Participants
  Acute kidney injury | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Allergic reaction | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Anorexia | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ascites | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Atrial fibrillation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Chills | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cough | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Decreased urine output | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dehydration | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dyspnea | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Edema | 2 | 1 | 0 | 6 | 2 | 1 | 0 | 3 | 4 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
  Electrolyte disturbances | 1 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Elevated LFT's | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Fatigue | 2 | 3 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Fever | 1 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Generalized pain | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GI disturbances | 2 | 0 | 0 | 6 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia | 4 | 6 | 0 | 7 | 7 | 0 | 0 | 4 | 6 | 1 | 0 | 3 | 0 | 0 | 2 | 4 | 2
  Hypocalcemia | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hyponatremia | 4 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypophosphatemia | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypotension | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 2
  Hypoxia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infusion-related reactions | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Myalgia | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea and vomiting | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Pericardial effusion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pleural effusion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pleuritic pain | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Proteinuria | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
  Pulmonary edema | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash and pruritis | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Tachycardia | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Ventricular dysfunction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Weight gain | 2 | 1 | 1 | 4 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 | Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
Number analyzed (Participants) | 6 | 8 | 6 | 6 | 3 | 6 | 5
Participants | 6 | 8 | 6 | 6 | 3 | 6 | 5

11. Other Pre Specified Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT)
Description: A DLT is defined per protocol as events attributed to LMB-100 and occurring during the DLT period such as hematological toxicities: Grade 4 neutropenia, Grade 3 and 4 febrile neutropenia, Grade 4 thrombocytopenia, and Grade 3 thrombocytopenia associated with bleeding episodes. Grade ≥3 non-hematological toxicity with the exception of: Grade 3 nausea and vomiting without appropriate treatment, Grade 3 diarrhea lasting ≤2 days with no fever or dehydration, and isolated Grade 3 fever. Grade ≥4 non-hematological toxicity: infusion related reactions, and any other drug related toxicity qualified as a DLT per the discretion of the principal investigator.
Time Frame: First 28 days following infusion of LMB-100 on Cycle 1, Day 1 through the duration of the study treatment up to 1 year.
Population: Arm A2 Phase 2 is not shown because it is not applicable due to dose expansion.
Measure: Count of Participants; unit: Participants
Groups:
- Arm B1, DL1, Phase I 48-hr Continuous Infusion Single Agent Lead-in: Arm B1, DL1, 48-hr Continuous Infusion Single Agent Lead-in 65µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered IV for 48 hours continuously on the first 1 - 4 days of each 21 day cycle for a maximum of 2 cycles
- Arm B1, DL3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in: Arm B1, DL3R, 24-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered IV for 24 hours continuously starting on days 1 and 4 of each 21 day cycle for a maximum of 2 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, DL1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, DL3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
Number analyzed (Participants) | 6 | 8 | 6 | 3 | 6 | 5
Participants
  Grade 3 Edema | 0 | 1 | 0 | 0 | 0 | 1
  Grade 3 Fatigue | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hypotension | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 Myalgia | 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 Urine output decreased | 0 | 1 | 0 | 0 | 0 | 1
  Grade 3 proteinuria | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 creatinine increase | 0 | 0 | 0 | 0 | 1 | 0

12. Other Pre Specified Outcome: Area Under the Plasma Concentration vs. Time Curve Extrapolated to Infinity (AUCinf)
Description: Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0). It is used to characterize drug absorption.
Time Frame: For Arms A1 & A2: Pre-dose, end of infusion (EOI), 1, 2 and 4 hours after EOI during Cycle 1 Day 1.
Population: Extended serum drug concentrations are available for all participants during Cycle 1. During Cycle 2, these bloods were not drawn (per protocol) after the first few participants on study, therefore elimination rate and AUC could only be calculated for Cycle 1 in most patients. Results from all participants receiving 65 mcg/kg short infusion were combined for the pharmacokinetic analysis as all received the same dose of LMB-100.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100: All participants in Arm A1 DL1.
- Arm A1 and Arm A2, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100: All participants in Arms A1 & A2, DL-1
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1 and Arm A2, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100
Number analyzed (Participants) | 6 | 14
h*ng/mL | 2,550 (38.2) | 1,409 (47.9)

13. Other Pre Specified Outcome: Area Under the Serum Concentration Versus Time Curve Extrapolated to Infinity (AUCinf)/D (Dose)
Description: The AUC is a measure of the serum concentration of the drug dose over time. It is used to characterize drug absorption.
Time Frame: For Arms A1 & A2: Pre-dose, end of infusion (EOI), 1, 2 and 4 hours after EOI during Cycle 1 Day 1.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: H*ng/mL/mg
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1 and Arm A2, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100
Number analyzed (Participants) | 6 | 14
H*ng/mL/mg | 415 (56.5) | 315 (45.8)

14. Other Pre Specified Outcome: Area Under the Serum Concentration Versus Time Curve Extrapolated to Last Measurement (AUClast)/D
Description: The AUC is a measure of the serum concentration of the drug dose over time. It is used to characterize drug absorption
Time Frame: For Arms B1 & B2: Pre-dose, end of loading dose, 2 and 6 hours after start of continuous infusion, end of infusion (EOI) and 2 hrs after EOI during Cycle 1 Day 1.
Population: Extended serum drug concentrations are avail. for all participants during C1. During C2, these bloods were not drawn (per protocol) after the first few participants on study, therefore elimination rate & AUC could only be calculated for C1 in most pts. AUClast is reported for Arms B1 and B2 as the measurements taken do not permit calculation of AUCinf.
Measure: Median (Standard Deviation); unit: h*ng/ml/mg
Arm/Group | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 5
h*ng/ml/mg | 519 (604) | 229 (71) | 233 (64) | 288 (184)

15. Other Pre Specified Outcome: Time Curve Extrapolated to Last Measurement (AUClast) for LMB-100
Description: Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated to last measurement. It is used to characterize drug absorption.
Time Frame: For Arms B1 & B2: Pre-dose, end of loading dose, 2 and 6 hours after start of continuous infusion, end of infusion (EOI) and 2 hrs after EOI during Cycle 1.
Population: Extended serum drug concentrations are avail. for all participants during C1. During C2, these bloods were not drawn (per protocol) after the first few participants on study, therefore elimination rate &AUC could only be calculated for C1 in most pts. AUClast is reported for Arms B1 and B2 as the measurements taken do not permit calculation of AUCinf.
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 5
h*ng/ml | 2671 (2778) | 4148 (1746) | 2508 (388) | 2417 (1006)

16. Other Pre Specified Outcome: The Total Clearance (CL) of LMB-100
Description: The CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: For Arms A1 & A2: Pre-dose, end of infusion (EOI), 1, 2 and 4 hours after EOI during Cycle 1 Day 1.
Population: LMB100 plasma conc. avail. for 20 pts on Arms A1/A2. Extended plasma drug conc. avail. for all pts during C1. During C2, these bloods were not drawn (per protocol) after1st few pts on study; elimination rate & T1/2 could only be calc. for C1 in most pts. Results from all pts w/65 mcg/kg short infusion were combined for the pharmacokinetic analysis (all rec'd same dose LMB-100). Arms B1/B2 calc. of T1/2 was not planned & plasma sample time points were inappropriate for computing this measure.
Measure: Mean (Standard Deviation); unit: L/h
Groups:
- Arms A1 & A2, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100: Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 Arm A1, DL1, Ph I Short Infusion 100µg/kg LMB-100 +125mg/m^2 nab-paclitaxel LMB-100 (short infusion): Administered intravenously (IV) on days 1, 3 and 5 of a 21 day cycle for a maximum of 2 cycles;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on days 1, and 8 of each 21 day cycle for a maximum of 2 cycles AND Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 Arm A1, DL-1, Ph I Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel LMB-100 (short infusion): Administered intravenously (IV) on days 1, 3 and 5 of a 21 day cycle for a maximum of 2 cycles;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on days 1, and 8 of each 21 day cycle for a maximum of 2 cycles AND Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 Arm A2, Ph 2 Short Infusion 65µg/kg LMB-100 +125mg/m^2 nab-paclitaxel LMB-100 (short infusion): Administered intravenously (IV) on days 1, 3 and 5 of a 21 day cycle for a maximum of 2 cycles;125mg/m^2 Nab-Paclitaxel: Administered intravenously (IV) on days 1, and 8 of each 21 day cycle for a maximum of 2 cycles
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arms A1 & A2, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100
Number analyzed (Participants) | 6 | 14
L/h | 2.97 (44.3) | 4.98 (116)

17. Other Pre Specified Outcome: Plasma Half-Life (T1/2) of LMB-100
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: For Arms A1 & A2: Pre-dose, end of infusion (EOI), 1, 2 and 4 hours after EOI during Cycle 1, Day 1.
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hour(h)
Groups:
- Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100: All participants in Arm A1, DL1.
- Arm A1 & A2, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100: All participants in Arm A1, DL-1 and Arm A2, DL-1.
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1 & A2, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100
Number analyzed (Participants) | 6 | 14
hour(h) | 1.25 (53.9) | 0.99 (12.9)

18. Other Pre Specified Outcome: Volume of Distribution (Vd) of LMB-100
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: For Arms A1 & A2: Pre-dose, end of infusion (EOI), 1, 2 and 4 hours after EOI during Cycle 1, Day 1.
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arms A1 & A2, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100
Number analyzed (Participants) | 6 | 14
L | 4.91 (20.5) | 7.48 (106)

19. Other Pre Specified Outcome: Maximum Observed (Peak) Plasma Concentration (Cmax) of LMB-100 in Arm A1 and Arm A2
Description: The maximum observed analyte concentration in serum was reported.
Time Frame: For Arms A1 & A2: Pre-dose, end of infusion (EOI), 1, 2 and 4 hours after EOI during Cycle 1 Day. Pre-dose and end of infusion (EOI) during Cycle 2 Day 1.
Population: LMB-100 peak plasma concentrations were available for all patients treated on study. Results from all participants receiving 65 mcg/kg short infusion (Arms A1 & A2) were combined for the pharmacokinetic analysis as all received the same dose of LMB-100.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Arms A1 & A2, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100: All participants in Arm A1, DL-1 and Arm A2.
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arms A1 & A2, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100
Number analyzed (Participants) | 6 | 14
ng/mL
  Cycle 1 Day 1 | 1,282 (14.9) | 858.9 (43.0)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 8
  Cycle 2 Day 1 | 1,306 | 748 (58.1)

20. Other Pre Specified Outcome: Maximum Observed (Peak) Plasma Concentration (Cmax) of LMB-100 in Arm B1 and Arm B2
Description: The maximum observed analyte concentration in serum was reported.
Time Frame: For Arms B1 & B2: Pre-dose, end of loading dose, 2 and 6 hours after start of continuous infusion, end of infusion (EOI) and 2 hrs after EOI during Cycle 1 Day 1. Pre-dose, end of loading dose and EOI during Cycle 2 Day 1.
Population: LMB-100 peak plasma concentrations were available for all patients treated on study. The Cmax reported for Arms B1 DL2 and DL3R and for Arm B2 occurred at end of the loading dose. Only non-zero values are reported for two participants in Cycle 2.
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 5
ng/mL
  Cycle 1 Day 1 | 1124 (1892) | 488 (270) | 485 (154) | 307 (163)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 3
  Cycle 2 Day 1 |  | 371 |  | 195 (248)

21. Other Pre Specified Outcome: Maximum Observed (Peak) Plasma Concentration (Cmax)/D (Dose) of LMB-100 in Arm A1 and Arm A2
Description: The maximum observed analyte concentration of dose was reported.
Time Frame: For Arms A1 & A2: Pre-dose, end of infusion (EOI), 1, 2 and 4 hours after EOI during Cycle 1 Day 1. Pre-dose and end of infusion (EOI) during Cycle 2 Day 1.
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Groups:
- Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100: All participants in Arm A1, DL-1 and Arm A2.
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100
Number analyzed (Participants) | 6 | 14
ng/mL/mg
  Cycle 1 Day 1 | 197 (18.5) | 188 (77.7)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 8
  Cycle 2 Day 1 | 181 | 158 (51.9)

22. Other Pre Specified Outcome: Maximum Observed (Peak) Plasma Concentration (Cmax)/D (Dose) of LMB-100 in Arm B1 and Arm B2
Description: The maximum observed analyte concentration in serum was reported.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1, Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 5
ng/mL
  Cycle 1 Day 1 | 235 (398) | 26.3 (12.1) | 45.1 (18.5) | 34.5 (19.8)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 3
  Cycle 2 Day 1 |  | 20.8 |  | 10.5 (5.9)

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 11 months, 8 days for A1DL1; 20 months, 9 days A1DL-1; 10 months, 17 days for A2; 2 months, 16 days for B1DL1; 14 months, 30 days for B1DL2; 5 months, 1 day for B2; and 4 months, 15 days for B1DL3R.
Groups:
- Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in 10: Arm B1, DL2, 48-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered intravenously (IV)for 48 hours continuously on the first 1 - 2 days of each 21 day cycle for a maximum of 2 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.
- Arm B1,Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in: Arm B1, DL3R, 24-hr Continuous Infusion Single Agent Lead-in 100µg/kg/day LMB-100 (continuous infusion LMB-100 as a single agent): Administered IV for 24 hours continuously starting on days 1 and 4 of each 21 day cycle for a maximum of 2 cycles. A 40 mcg/kg loading dose of LMB-100 is administered over 30 minutes immediately prior to the start of each long infusion.
Arm/Group | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 | Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in 10 | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in | Arm B1,Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg
All-Cause Mortality (participants affected / at risk) | 5/6 | 8/8 | 5/6 | 6/6 | 3/3 | 6/6 | 3/5
Serious Adverse Events (participants affected / at risk) | 3/6 | 4/8 | 1/6 | 2/6 | 2/3 | 2/6 | 1/5
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 6/6 | 6/6 | 3/3 | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 (N=6) | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 (N=8) | Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 (N=6) | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in 10 (N=6) | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in (N=3) | Arm B1,Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in (N=6) | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg (N=5)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, died at home (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A1, Dose Level 1, Phase I Short Infusion 100µg/kg LMB-100 (N=6) | Arm A1, Dose Level-1, Phase I Short Infusion 65µg/kg LMB-100 (N=8) | Arm A2, Phase 2 Short Infusion 65µg/kg LMB-100 (N=6) | Arm B1, Dose Level 2, Phase I 48-hr Continuous Infusion Single Agent Lead-in 10 (N=6) | Arm B1, Dose Level 1, Phase I 48-hr Continuous Infusion Single Agent Lead-in (N=3) | Arm B1,Dose Level 3R, Phase I 24-hr Continuous Infusion Single Agent Lead-in (N=6) | Arm B2, Phase I 24-hr Continuous Infusion Combo Therapy 100µg/kg (N=5)
Platelet count decreased (Investigations) | 1 (2) | 4 (4) | 3 (3) | 2 (3) | 2 (4) | 2 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, tachypnea intermittent (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (7) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Skin and subcutaneous tissue disorders - Other, buttock excoriation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 2 (6) | 4 (6) | 3 (10) | 2 (8) | 1 (3) | 1 (2) | 2 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 4 (12) | 6 (18) | 4 (7) | 0 (0) | 0 (0) | 1 (2) | 3 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (6):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT02810418/Prot_SAP_000.pdf
  • Informed Consent Form: Screening Consent (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02810418/ICF_001.pdf
  • Informed Consent Form: Arm A1 Phase I Short Infusion Consent (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02810418/ICF_002.pdf
  • Informed Consent Form: Arm A2 Phase II Short Infusion Consent (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02810418/ICF_003.pdf
  • Informed Consent Form: Arm B1 Continuous Infusion Single Agent (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02810418/ICF_004.pdf
  • Informed Consent Form: Arm B2 Continuous Infusion Combo Consent (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02810418/ICF_005.pdf